CLINICAL TRIAL: NCT02609750
Title: WorkUp. Early Structured Care Including Workplace Interventions to Improve Work Ability in Patients With Neck and/or Back Pain. A Prospective Pare Wise Cluster Randomized Controlled Trial in Primary Care With One Year Follow up
Brief Title: WorkUp. Structured Care With Workplace Interventions to Improve Work Ability in Patients With Neck and/or Low Back Pain
Acronym: WorkUp
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other); Kronoberg County Council (Other Government); Blekinge County Council Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS2011/005
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Back Pain; Neck Pain
MeSH Terms: conditions — Back Pain; Neck Pain | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured care & workplace intervention (Experimental): Through a flow chart the investigators in detail specify the medical and work place interventions (all according to evidence-based guidelines). Red, yellow and blue flags, and motivational factors are identified in a screening investigation. The aim of the screening is to individually tailor the rehabilitation interventions. Physiotherapy interventions are based on a bio-psychosocial and cognitive behavioural therapy perspective. Behavioural medicine treatment principles include careful examination and treatments such as advice to stay active, instructions, OMI, OMT, MDT. The investigators apply interventions based on ergonomics, motivational factors and work place changes according to Convergence Dialogue Meetings (CDM).
  Interventions: Other: Structured care & workplace intervention
- Treatment as Usual (Active Comparator): Patients follows the PHCs standard schedule and procedures including the so called rehabilitation guarantee
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Structured care & workplace intervention — In addition to structured care a workplace intervention named Convergence Dialogue Meetings (CDM) are carried out. CDM is a three step structured dialogue and meeting model supporting the patient, health care professionals and employer to summarize concrete suggestions to support sustainable work ability and a return to work if sick listed.
  Arms: Structured care & workplace intervention
Other: Treatment as Usual — Patients will follow the primary health care's standard time schedule and procedures as of ordinary care and the rehabilitation guarantee. For each patient all treatment measures are recorded in a manual, regarding number of treatments, time used per treatment and type of treatment.
  Arms: Treatment as Usual

SUMMARY:
WorkUp is a prospective cluster randomised controlled trial in primary care. The main purpose is to investigate effects of early structured care based on screening of red flags (signs of serious medical conditions/disease), yellow flags (psychosocial factors, attitude to pain) and blue flags (workplace related factors) and including a workplace intervention according to the method "Convergence Dialogue Meetings" (CDM) for improving work ability, in comparison with treatment as usual, in patients with neck and/or back pain.

DETAILED DESCRIPTION:
Musculoskeletal disorders are the most common reasons for sick leave in western countries. Identifying risk factors and predictors for a stable return to work (RTW ) is essential. An evidence-based safe care includes systems for detecting medical conditions with urgent need for care (red flags) and psycho-social risk factors (yellow flags). To maintain work ability, also requires different capacities related to work demands, (physical, mental and social) as well as work environment aspects covered by a "blue flag system".

Since motivation is assumed to drive and sustain human behaviour, patients with back pain seek health care when motivation reaches a threshold level. Patients want to be examined, get treatment and self-care advice to resume normal daily activities. This might lead to improved long-standing results in terms of health, function and work ability.

The investigators hypothesize that WorkUp, a timely tailor-made and evidence-based intervention leads to a faster recovery of health, function and RTW as compared to standard care. This includes the identification of both the patient's risk factors (red, yellow and blue flags) and motivational factors. Based on this screening, a structured tailored intervention will be offered. The WorkUp model comprise of evidence-based treatment and interaction between patient, health care and work place interventions.

The main purpose is to test WorkUp in a comparison study with treatment as usual (TAU) in primary health care (PHC).

Design: A prospective paire wise cluster randomized trial in PHC including a one year clinical follow-up and a three year register follow-up.

Intervention: Through a flow chart the investigators in detail specify the medical and work place interventions (all according to evidence-based guidelines). Red, yellow and blue flags, and motivational factors are identified in a screening investigation. The aim of the screening is to individually tailor the rehabilitation interventions. Physiotherapy interventions are based on a bio-psychosocial and cognitive behavioural therapy perspective. Behavioural medicine treatment principles will include careful examination and treatments such as advice to stay active, instructions, OMI, OMT, MDT. The investigators apply interventions based on ergonomics, motivational factors and work place changes according to Convergence Dialogue Meetings(CDM). CDM is a three step structured dialogue and meeting model supporting the patient, health care professionals and employer to summarize concrete suggestions to support a RTW .

TAU patients follow the PHC's standard schedule and procedures including the so called rehabilitation guarantee.

For each patient all treatment measures are recorded in a protocol.

A power analysis indicated that the investigators needed to recruit a minimum of 20 PHCs and 500 patients.

This type of structured routine primary care can facilitate an adequate treatment for patients with musculoskeletal pain and how to allocate sparse resources. If beneficial results emerge a structured implementation program will follow.

ELIGIBILITY:
Inclusion Criteria:

* acute and subacute neck and/or back pain (less than three months of duration)
* a working history of at least four weeks during the last year
* being at risk for sick leave according to the short form of the Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ) (cut off >40)
* if sickness absent < 60 days.

Exclusion Criteria:

* identified abuse
* retirement pension
* ongoing acute medical treatment
* pregnancy

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Work ability | Changes from baseline to after treatment (3, 6, 12 months and 2 and 3 years)
  Work ability (defined as being at work or being eligible to the labour market during at least four weeks in a row) and time of sickness absence and Return to work. Year 2 and 3 follow-up by register data

SECONDARY OUTCOMES:
Health-related quality of life | Changes from baseline to after treatment (3, 6 and 12 months)
  Measured by EQ-5D (Euroqol 2011 EQ-5D)
Functional ability | Changes from baseline to after treatment (3, 6 and 12 months)
  Measured by the Oswestry Disability Index (ODI) in low back pain patients (Fairbank & Pynsent 2000) and by the Neck Disability Index (NDI) in patients with neck pain (MacDermid et al 2009)
Pain (distribution and intensity) | Changes from baseline to after treatment (3, 6 and 12 months)
  Measured by the Pain mannequin (Bergman et al 2001) and VAS (Sieper et al 2009)
Physical and psycho-social work environment | Changes from baseline to after treatment (3, 6 and 12 months)
  Measured by questions focusing on known risk factors according to Lindell´s thesis (2010) and the ULF questionnaire
Patient´s satisfaction | Changes from baseline to after treatemnt (3, 6 and 12 months)
  Measured by use of the Client Satisfaction Questionnaire (CSQ) (Bjelland 2002)

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta EM Grahn, AssProfessor, Principal Investigator — Dep of Clinical Sciences Lund, Orthopedics, Lund University, and FoU Kronoberg, Region Kronoberg

REFERENCES:
- [Derived] Axen I, Sennehed CP, Eek F, Stigmar K. Can a workplace dialogue impact the perceived influence of neck and/or backpain on everyday activities and performance at work? A secondary analysis from the randomized controlled trial WorkUp. BMC Musculoskelet Disord. 2022 Sep 15;23(1):861. doi: 10.1186/s12891-022-05812-w. PMID 36104781
- [Derived] Forsbrand MH, Turkiewicz A, Petersson IF, Sennehed CP, Stigmar K. Long-term effects on function, health-related quality of life and work ability after structured physiotherapy including a workplace intervention. A secondary analysis of a randomised controlled trial (WorkUp) in primary care for patients with neck and/or back pain. Scand J Prim Health Care. 2020 Mar;38(1):92-100. doi: 10.1080/02813432.2020.1717081. Epub 2020 Jan 30. PMID 32000558
- [Derived] Forsbrand MH, Grahn B, Hill JC, Petersson IF, Post Sennehed C, Stigmar K. Can the STarT Back Tool predict health-related quality of life and work ability after an acute/subacute episode with back or neck pain? A psychometric validation study in primary care. BMJ Open. 2018 Dec 22;8(12):e021748. doi: 10.1136/bmjopen-2018-021748. PMID 30580256
- [Derived] Saha S, Grahn B, Gerdtham UG, Stigmar K, Holmberg S, Jarl J. Structured physiotherapy including a work place intervention for patients with neck and/or back pain in primary care: an economic evaluation. Eur J Health Econ. 2019 Mar;20(2):317-327. doi: 10.1007/s10198-018-1003-1. Epub 2018 Aug 31. PMID 30171489
- [Derived] Sennehed CP, Holmberg S, Axen I, Stigmar K, Forsbrand M, Petersson IF, Grahn B. Early workplace dialogue in physiotherapy practice improved work ability at 1-year follow-up-WorkUp, a randomised controlled trial in primary care. Pain. 2018 Aug;159(8):1456-1464. doi: 10.1097/j.pain.0000000000001216. PMID 29554017
- [Derived] Forsbrand M, Grahn B, Hill JC, Petersson IF, Sennehed CP, Stigmar K. Comparison of the Swedish STarT Back Screening Tool and the Short Form of the Orebro Musculoskeletal Pain Screening Questionnaire in patients with acute or subacute back and neck pain. BMC Musculoskelet Disord. 2017 Feb 21;18(1):89. doi: 10.1186/s12891-017-1449-9. PMID 28222707